CLINICAL TRIAL: NCT06329141
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Groups, Phase 2a Clinical Trial to Assess the Efficacy and Safety of Vutiglabridin in Early Parkinson's Disease Patients
Brief Title: A Study to Assess the Efficacy and Safety of Vutiglabridin in Early Parkinson's Disease Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Glaceum (Industry)
Collaborators: The Catholic University of Korea (Other); Kyunghee University Medical Center (Other); Korea University Guro Hospital (Other); Samsung Medical Center (Other); Severance Hospital (Other); Inje University (Other); Hallym University Medical Center (Other); The Catholic University of Korea Uijeongbu St.Marys Hostpial (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSG4112-P2-03
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Vutiglabridin 400 mg Multiple Dose (Experimental): Multiple oral dosing of vutiglabridin 400 mg for 24 weeks
  Interventions: Drug: Vutiglabridin
- Vutiglabridin 800 mg Multiple Dose (Experimental): Multiple oral dosing of vutiglabridin 800 mg for 24 weeks
  Interventions: Drug: Vutiglabridin
- Placebo (Placebo Comparator): Multiple oral dosing of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vutiglabridin — Once-daily oral administration
  Other Names: HSG4112; 2-(8,8 dimethyl 2,3,4,8,9,10 hexahydropyrano[2,3 f]chromen 3 yl) 5 ethoxyphenol
  Arms: Vutiglabridin 400 mg Multiple Dose; Vutiglabridin 800 mg Multiple Dose
Drug: Placebo — Once-daily oral administration
  Arms: Placebo

SUMMARY:
1. Study Objective

   - To assess the efficacy and safety of vutiglabridin in early Parkindson's disease patients
2. Background Glaceum Inc. has evaluated the safety, tolerability, and pharmacokinetic/pharmacodynamic properties of vutiglabridin in healthy subjects through its Phase 1 trials, and is planning to perform this Phase 2a trial to assess the efficacy and safety of vutiglabridin in early Parkinson's disease patients.
3. Study Design and Protocol This study is a randomized, double-blind, placebo-controlled, parallel-group trial. Subjects deemed eligible to participate in this study based on the inclusion/exclusion criteria will be assigned a subject number and randomized to one of the 3 treatment groups - 1 group receiving a placebo - in a 1:1:1 ratio. Subjects will be randomized to double-blind treatments and will receive a once-daily oral dose of the investigational product for 24 weeks according to the study protocol. Several parameters (i.e., MDS-UPDRS, CGI-C, K-NMSS, modified Hoehn-Yahr stage and SNBR) will be evaluated to assess the efficacy of vutiglabridin. Assessments including measurement of vital signs, 12-lead ECG, clinical laboratory test, pregnancy test, physical examination, and adverse event monitoring will be performed to evaluate the safety and tolerability of vutiglabridin. Blood samples will be collected for pharmacokinetic assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand, and provide written consent for the trial, comply with the clinical trial protocol, and communicate any adverse events (AEs) and other clinically significant information to the investigator (able to complete the evaluation, including walking or using walking aids).
2. Adult men and women between the ages of 40 and 75 at Screening.
3. Diagnosed with Parkinson's disease according to the UK Parkinson's Disease Society (UKPDS) Brain Bank clinical diagnostic criteria and confirmed the reduction of dopamine transporter on 18F-FP-CIT PET imaging at Screening.
4. Diagnosed with Parkinson's disease within the last 24 months.
5. Hoehn-Yahr stage ≤ 2
6. Eligible females will be:

   * females of childbearing potential who are not pregnant, evidenced by a negative serum hCG pregnancy test at Screening
   * non-lactating, or
   * surgically sterile (defined as documented bilateral tubal ligation, bilateral tubal occlusion, bilateral oophorectomy, hysterectomy) or postmenopausal.

     * Definition of menopause
   * 50 years or over: 12 or more consecutive months without menstruation, in the absence of other conditions.
   * Less than 50 years: FSH level is > 40 IU/L and 12 or more consecutive months without menstruation, in the absence of other conditions.

Exclusion Criteria:

1. Clinically significant new illness, per Investigator judgment, in the 4 weeks before Screening and during the screening period.
2. Global Deterioration Scale (GDS) ≥ 4 at Screening.
3. Have clinically significant depression as indicated by a Korean Beck Depression Inventory II score (K-BDI-II) > 18 at Screening.
4. BMI less than 18.5 kg/m2 at Screening.
5. Have the following laboratory test results:

   * Clinically significant abnormal hepatic (i.e., AST or ALT greater than 2.5x ULN, or total bilirubin greater than 2x ULN, unless documented Gilbert's syndrome)
   * Renal function laboratory test (i.e., GFR < 60 mL/min).
6. Have the following medical history:

   * Diagnosed with or suspected to have *Parkinson-plus syndromes (PPS)

     * PPS: Multiple System Atrophy, Progressive Supranuclear Palsy, Corticobasal Degeneration, Diffuse Lewy Body Disease, etc.
   * Tremor-dominant Parkinson's disease, per Investigator judgment.
   * Symptoms or signs indicative of neurological functional impairment or known abnormalities in brain CT or MRI imaging.
   * A history of severe heart failure (NYHA class III ~ IV), stroke, cerebral ischemic attacks, or seizures within the past year before screening; or those with a history of myocardial infarction or unstable angina within the last 6 months before screening.
   * Have undergone surgery for Parkinson's disease treatment (e.g., cholecystectomy, deep brain stimulation, fetal tissue transplantation) or any other major brain surgery.
   * Diagnosed with malignant tumors within the past 5 years before screening (except for adequately treated basal cell carcinoma, cervical intraepithelial neoplasia, thyroid cancer, or flat epithelial atypia).
   * Diagnosed with secondary Parkinsonism (drug-induced Parkinsonism, normal pressure hydrocephalus, vascular Parkinsonism).
7. Have swallowing problems
8. Have clinically significant dizziness, nausea, per Investigator's judgment.
9. Currently taking any of the following medications and have the willingness and ability to continue taking them throughout the clinical trial period:

   * Within the 4 weeks before baseline, taking any Parkinson's disease medications, including dopamine agonists, dopamine-depleting enzyme inhibitors [monoamine oxidase inhibitors (MAOi), COMT (catechol-O-methyltransferase) inhibitors], non-dopaminergic drugs (anticholinergic agents, amantadine, etc.), and others PD medications (In case of irreversible MAO-B inhibitor, within the 90 days before baseline)
   * Within the 12 weeks before screening, have used systemic steroids continuously for 7 days or longer.
   * Within the 12 weeks before baseline, taking levodopa or levodopa combinations (except history of levodopa use for more than 4 weeks)
   * Currently taking medications known to be substrates of breast cancer resistant protein (BCRP) at screening (e.g., rosuvastatin, serpalan, etc.) (Note: If switched to another drug of the same class, the subject may be eligible for inclusion).
   * taking of any medication within 6 months of Screening that can alter reproductive hormone levels, either as the intended effect or as a side effect, including: anabolic steroids, androstenedione, bicalutamide, cimetidine, dehydroepiandrosterone, diethylstilbestrol, other estrogens, dutasteride, finasteride, glucocorticoids (e.g., prednisone, cortisone, hydrocortisone, and decadron), oral ketoconazole, megestrol acetate, opiates (e.g., morphine, codeine, oxycodone, hydrocodone), spironolactone, testosterone or any androgen, and any medications for treating prostate cancer.
10. Have taken of stable doses of levodopa or levodopa combination
11. Have known or suspected intolerance to PET scan or fluoropropyl-CIT (18F).
12. Have a history of organ transplantation.
13. Tested positive for HBsAg, HCV Ab, HIV Ag/Ab, or VDRL(RPR) antibodies in screening tests.
14. Known hypersensitivity or contraindication to the main ingredient and excipients of the investigational product.
15. Anticipated to undergo surgery during the clinical trial period or to receive surgical interventions that may affect the completion of the trial or compliance with the clinical trial protocol.
16. Participated in a clinical trial for an investigational drug or medical device for a period equal to or longer than five times the drug's half-life at baseline or within the past 12 weeks, whichever is longer.
17. Unwilling, or whose partner is unwilling, to use a medically acceptable means of *contraception during and for 90 days following completion/withdrawal of the study.

    * Medically acceptable contraceptive methods include:

      * intrauterine device that has been proven highly effective, used by the subject or the subject's spouse/partner
      * physical contraception (male or female) used with chemical sterilization surgical sterilization of the subject or the subject's partner (e.g., vasectomy, hysterectomy, tubal ligation, salpingectomy
      * oral hormonal contraceptive used by the spouse/partner of male subject.
18. Within the last 2 years before screening or during the screening period, have a history of alcohol or drug abuse, or have tested positive for drug use during the screening period (Note: Subjects who have used drugs for the purpose of chronic pain treatment, have documented records of medical history and concomitant medications, may, at the investigator's discretion and with the sponsor's approval, be eligible for inclusion as trial subjects).
19. Deemed unsuitable for participation in the clinical trial by the investigator due to reasons including clinical laboratory test results and other factors.
20. Participating in a non-interventional clinical study that may affect the safety or efficacy assessment of subjects in this clinical trial.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in MDS-UPDRS Part III Subscore | From baseline to Week 24

SECONDARY OUTCOMES:
Change From Baseline in MDS-UPDRS Part III Subscore | From baseline to Week 4, Week 12, Week 28
Change From Baseline in MDS-UPDRS Part II + Part III | From baseline to Week 4, Week 12, Week 28
Change From Baseline in CGI-C score | From baseline to Week 4, Week 12, Week 24
Change From Baseline in K-NMSS score | From baseline to Week 4, Week 24
Change From Baseline in Modified Hoehn-Yahr stage | From baseline to Week 4, Week 12, Week 24
Change From Baseline in PET SNBR (Specific to Non-specific Binding Ratio) in the putamen, acudate and nucleus | From baseline to Week 24
Drop-out rate due to taking anti-parkinson drug | From baseline to Week 28 (follow-up visit)

CONTACTS AND LOCATIONS:
Locations (9):
- South Korea (9):
  - Hallym University Medical Center, Anyang-si, Gyeonggi-do
  - The Catholic University of Korea Uijeongbu St.Marys Hostpial, Uijeongbu-si, Gyeonggi-do
  - Inje University Busan Paik Hospital, Busan
  - Inje University Sanggye Paik Hospital, Seoul
  - KyungHee University Medical Center, Seoul
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul
  - Korea University Guro Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No